CLINICAL TRIAL: NCT03021122
Title: Reducing Medication Errors and Time to Vasoactive Drugs Preparation and Delivery During Pediatric Cardiopulmonary Resuscitation: a Multicenter, Prospective, Randomized Controlled Trial
Brief Title: Reducing Medication Errors and Time to Drugs Delivery During Pediatric Cardiopulmonary Resuscitation: a Multicenter RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pediatric Clinical Research Platform (Other)
Collaborators: University of Geneva, Switzerland (Other); University of Lausanne Hospitals (Other); Insel Gruppe AG, University Hospital Bern (Other); Neuchâtel Hospital, Neuchâtel, Switzerland (Unknown); Fribourg Hospital, Fribourg, Switzerland (Unknown); Sion Hospital, Sion, Switzerland (Unknown)
Responsible Party: Principal Investigator, Johan Siebert, MD: Emergency Physician, University Hospital, Geneva
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SNSF_32003B_169348
Record Dates: First submitted 2017-01-12; First posted 2017-01-13 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Resuscitation; Pediatrics
Keywords: Medication errors; Resuscitation; Drugs; Pediatrics; Biomedical technology

STUDY DESIGN:
Who Masked: Participant
Masking Description: Blinding to the purpose of the study during recruitment will be maintained to minimize preparation bias. Nurses will be "unblinded" when the simulated scenario start.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (PedAMINES™ / Conventional Method) (Experimental): A 2-period study where nurses will be randomized to a 15-minute CPR scenario to prepare and deliver Dopamine with the help of PedAMINES™ first, then crossover (incl. washout period) to prepare and deliver Norepinephrine with the help of a Conventional Method.
  Interventions: Device: PedAMINES™ / Conventional Method
- Arm B (Conventional Method / PedAMINES™) (Active Comparator): A 2-period study where nurses will be randomized to a 15-minute CPR scenario to prepare and deliver Dopamine with the help of a Conventional Method first, then crossover (incl. washout period) to prepare and deliver Norepinephrine with the help of PedAMINES™.
  Interventions: Device: Conventional Method / PedAMINES™

INTERVENTIONS:
Device: PedAMINES™ / Conventional Method — Each nurse will be asked to prepare a 5 μg/kg/min continuous infusion of dopamine (Period 1) and then to prepare a 0.1 μg/kg/min continuous infusion of norepinephrine (Period 2) for a 25kg boy using the studied delivery devices according to the sequence randomly assigned based on a cross-over design:
  • PedAMINES™ (Period 1) and then Conventional Method (Period 2)
  Arms: Arm A (PedAMINES™ / Conventional Method)
Device: Conventional Method / PedAMINES™ — Each nurse will be asked to prepare a 5 μg/kg/min continuous infusion of dopamine (Period 1) and then to prepare a 0.1 μg/kg/min continuous infusion of norepinephrine (Period 2) for a 25kg boy using the studied delivery devices according to the sequence randomly assigned based on a cross-over design:
  • Conventional Method (Period 1) and then PedAMINES™ (Period 2)
  Arms: Arm B (Conventional Method / PedAMINES™)

SUMMARY:
The investigators recruit nurses working in 5 swiss Pediatric Emergency Departments or divisions to prepare continuous infusions of vasoactive drugs during a simulation-based pediatric CPR cardiac arrest scenario. According to randomization, nurses will have to prepare and deliver vasoactive drugs following their current conventional methods or by the aim of a mobile tablet application called PedAMINES™. PedAMINES™ is designed to support them step-by-step from order to delivery of these drugs.

1. Primary outcome will be to measure in each allocation group the number of medication dosage errors committed during each drug preparation sequence until injection.
2. Secondary outcome will be to measure the time to drug preparation (TDP) and time to drug delivery (TDD).

DETAILED DESCRIPTION:
During pediatric cardiopulmonary resuscitation (CPR), vasoactive drug preparation for continuous infusion is both complex and time-consuming, placing children at higher risk than adults for medication errors. It is well established that CPR duration is inversely correlated to survival, decreasing linearly by 2.1 % per minute, and to decreased risk of neurological sequelae [1].

In this study, the investigators recruit nurses working in 5 swiss Pediatric Emergency Departments or divisions to prepare continuous infusions of vasoactive drugs during a simulation-based pediatric CPR cardiac arrest scenario with a high-fidelity manikin (Laerdal SimJunior™). The scenario will take place in the shock room to increase realism.

According to randomization with a 1:1 allocation ratio, nurses will have to prepare and deliver vasoactive drugs following their current conventional methods or by the aim of a mobile tablet application called PedAMINES™ (Pediatric Accurate Medication In Emergency Situations). PedAMINES™ is designed to support nurses step-by-step from order to delivery of a wide range of drugs, especially those requiring continuous infusion. PedAMINES™ has already been shown in a single-center simulation-based study to reduce time to vasoactive drug preparation, to delivery and the rate of medication errors [2].

On the day of participation, after obtaining nurse's written informed consent and randomization, nurses will receive a standardized 5-minute training session on how to use the app. Then, the nurses will be asked to perform a standardized 15-minute highly realistic CPR scenario, including post-return of spontaneous circulation (ROSC). After epinephrine-induced ROSC, nurses will be asked to first prepare a continuous infusion of dopamine, using either PedAMINES™ or a conventional method, and then a continuous infusion of norepinephrine by crossing the procedure. Moreover, 2 questionnaires will be given before and after the scenario to ask the nurses about their demographics data, perceived stress and degree of satisfaction.

1. Primary outcome will be to measure in each allocation group the number of medication dosage errors committed during each drug preparation sequence until injection.
2. Secondary outcome will be to measure the time to drug preparation (TDP) and time to drug delivery (TDD).

All the actions (i.e. primary and secondary outcomes) performed by the nurses during the scenario will be automatically recorded and stored by the responsive simulator detectors, the application and by several video cameras. To avoid assessment bias, two evaluators will then independently review these video recordings. In case of disagreement, a third independent evaluator will help reach a consensus.

We aim to determine whether the use of PedAMINES™ might improve the management of acute life-threatening conditions by quickly delivering expertise in vasoactive drugs administration in other hospitals in Switzerland, even in non-university hospitals where nurses (and physicians) are either little or not exposed to pediatric CPRs. We hypothesize that PedAMINES™ might primary reduce medication errors, and secondary reduce delays to drugs preparation and delivery independently of the existing conventional preparation methods or nurses' skills.

ELIGIBILITY:
Inclusion Criteria:

* To be nurse certified
* To know how to prepare intravenous drugs injection.
* To have previously completed the 5-minute introductory course to the use of PedAMINES dispensed by the investigators of the study.
* Participation agreement

Exclusion Criteria:

* To have at any time undergone a previous experiment with a cognitive numeric device aimed to help vasoactive drugs preparation.
* To have not undergone the 5-minute introductory course to the use of PedAMINES.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Medication dosage errors | On the day of study participation
  To measure in each allocation group the number of medication dosage errors committed during each drug preparation sequence until injection.

SECONDARY OUTCOMES:
Time to drug preparation (TDP) and time to drug delivery (TDD) | On the day of study participation
  To measure in each allocation group the elapsed time in seconds between the oral prescription by the physician to drug preparation completion by the nurse (TDP) and to drug delivery (TDD) by the nurse.

CONTACTS AND LOCATIONS:
Overall Officials: Johan N Siebert, MD, Principal Investigator — Geneva Children Hospital, Geneva University Hospitals, Geneva, Switzerland
Locations (6):
- Switzerland (6):
  - Hôpital de l'Enfance (HEL), Lausanne, Canton of Vaud
  - Hôpital du Valais, Sion, Valais
  - Inselspital Bern, Bern
  - HFR Fribourg, Fribourg
  - Geneva Children's Hospital, Geneva University Hospitals, Geneva
  - Hôpital Neuchâtelois, Neuchâtel

IPD SHARING:
Plan to Share IPD: Yes
IPD will be deidentified and the study investigators will house the data locally on secure hard disk drives (HDD) at the Geneva Children's Hospital. Data will be freely available to anyone upon request 1 year after study completion. Only deidentified/anonymized data will be shared.

REFERENCES:
- [Background] Matos RI, Watson RS, Nadkarni VM, Huang HH, Berg RA, Meaney PA, Carroll CL, Berens RJ, Praestgaard A, Weissfeld L, Spinella PC; American Heart Association's Get With The Guidelines-Resuscitation (Formerly the National Registry of Cardiopulmonary Resuscitation) Investigators. Duration of cardiopulmonary resuscitation and illness category impact survival and neurologic outcomes for in-hospital pediatric cardiac arrests. Circulation. 2013 Jan 29;127(4):442-51. doi: 10.1161/CIRCULATIONAHA.112.125625. Epub 2013 Jan 22. PMID 23339874
- [Background] Siebert JN, Ehrler F, Combescure C, Lacroix L, Haddad K, Sanchez O, Gervaix A, Lovis C, Manzano S. A Mobile Device App to Reduce Time to Drug Delivery and Medication Errors During Simulated Pediatric Cardiopulmonary Resuscitation: A Randomized Controlled Trial. J Med Internet Res. 2017 Feb 1;19(2):e31. doi: 10.2196/jmir.7005. PMID 28148473
- [Derived] Siebert JN, Gosetto L, Sauvage M, Bloudeau L, Suppan L, Rodieux F, Haddad K, Hugon F, Gervaix A, Lovis C, Combescure C, Manzano S, Ehrler F; PedAMINES Trial Group; PedAMINES Prehospital Group. Usability Testing and Technology Acceptance of an mHealth App at the Point of Care During Simulated Pediatric In- and Out-of-Hospital Cardiopulmonary Resuscitations: Study Nested Within 2 Multicenter Randomized Controlled Trials. JMIR Hum Factors. 2022 Mar 1;9(1):e35399. doi: 10.2196/35399. PMID 35230243
- [Derived] Siebert JN, Ehrler F, Combescure C, Lovis C, Haddad K, Hugon F, Luterbacher F, Lacroix L, Gervaix A, Manzano S; PedAMINES Trial Group. A mobile device application to reduce medication errors and time to drug delivery during simulated paediatric cardiopulmonary resuscitation: a multicentre, randomised, controlled, crossover trial. Lancet Child Adolesc Health. 2019 May;3(5):303-311. doi: 10.1016/S2352-4642(19)30003-3. Epub 2019 Feb 21. PMID 30797722
- [Derived] Siebert JN, Ehrler F, Lovis C, Combescure C, Haddad K, Gervaix A, Manzano S. A Mobile Device App to Reduce Medication Errors and Time to Drug Delivery During Pediatric Cardiopulmonary Resuscitation: Study Protocol of a Multicenter Randomized Controlled Crossover Trial. JMIR Res Protoc. 2017 Aug 22;6(8):e167. doi: 10.2196/resprot.7901. PMID 28830854